CLINICAL TRIAL: NCT06129331
Title: Aortic Stenosis and Cardiac Amyloidosis: A Pragmatic, Streamlined International
Brief Title: Aortic Stenosis and Cardiac Amyloidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Allina Health System (Other); Royal Free Hospital NHS Foundation Trust (Other); Columbia University (Other); Medical University of South Carolina (Other); Laval University (Other); Vilnius University Hospital Santaros Klinikos (Other); Université Catholique de Louvain (Other); Wolfson Medical Center (Other Government); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Trieste (Other)
Responsible Party: Principal Investigator, Christian Nitsche, Principle Investigator, Medical University of Vienna
Other Study IDs: 2218_2016
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Amyloidosis; Aortic Stenosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AS-CA without amyloid-specific treatment: Patients with no amyloid-specific treatment
  Interventions: Other: No amyloid-specific treatment
- AS-CA with amyloid-specific treatment: Patients receiving newly available amyloid-specific drugs
  Interventions: Drug: Amyloid-specific treatment

INTERVENTIONS:
Drug: Amyloid-specific treatment — Amyloid-specific treatment
  Groups: AS-CA with amyloid-specific treatment
Other: No amyloid-specific treatment — No amyloid-specific treatment
  Groups: AS-CA without amyloid-specific treatment

SUMMARY:
The dual pathology of aortic stenosis (AS) and cardiac amyloidosis (CA) is increasingly recognized. Even tough efforts have been undertaken to bring cohorts together, the largest cohort of AS-ATTR to date is <50 patients. It is the aim of the present international, multi-center registry to collect ~300 patients with AS-CA creating a big enough cohort to allow

1. thorough characterization of this condition
2. assessment of log-term clinical outcomes of AS-CA
3. assessment of effectiveness of amyloid-specific treatment on top of valve replacement

DETAILED DESCRIPTION:
Calcific aortic stenosis (AS) and transthyretin (ATTR) cardiac amyloidosis are both conditions commonly affecting the elderly. Bone scintigraphy using amyloid-avid tracers (99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid, DPD; 99mTc-pyrophosphate; or 99mTc-hydroxymethylene diphosphonate) represents the key imaging modality for non-invasive ATTR diagnosis. Recent studies have used this technology to screen AS patients and demonstrated that AS and ATTR may coexist in 8 to 16%. This is substantially higher than in non-cardiac referrals for bone scintigraphy (range 1-3% in individuals >80 years), which is considered the most accurate approach to estimate the ATTR prevalence in the general population. While the dual burden of AS and ATTR might suggest adverse prognostic implications, it has been shown that AS-ATTR and lone AS patients benefit equally from transcatheter aortic valve replacement (TAVR) with comparable 1- and 2-year survival rates. Yet, data on long-term outcomes are still missing.

With increased recognition and valvular treatment of AS-ATTR, the disease course after TAVR becomes a key issue. Our data suggest significantly different remodeling between lone AS and AS-ATTR, with the latter being transformed into a "lone-ATTR" cardiomyopathy phenotype at one-year post-TAVR. Novel ATTR-specific treatments are now available, with the potential to further improve prognosis in AS-ATTR on top of valvular replacement. However, patients with significant AS were not included in the ATTR-ACT trial, and treatment effectiveness in this patient population therefore remains unclear. Also, despite increased ATTR screening globally, the case numbers for dual AS-ATTR of individual centers are still low.

The present international multi-center study is therefore designed to provide detailed characterization of dual AS-ATTR, inform about long-term clinical outcomes and assess the effect of ATTR specific treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant AS and a concomitant diagnosis of cardiac amyloidosis who are eligible for inclusion as per local permissions

Exclusion Criteria:

* Patients without significant AS (less than moderate AS)
* Patients with other subtypes of cardiac amyloidosis (e.g., light chain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a dual pathology of significant aortic stenosis and concomitant cardiac amyloidosis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Phenotyping of AS with "early" ATTR infiltration (DPD grade 1) versus "advanced" ATTR cardiomyopathy (DPD grade 2/3) | 0 months
  Dual pathology patients with DPD grade 1 will be compared to those with DPD grade 2/3 with regards to symptoms (New York Heart Association functional class), functional capacity (6-Minute walk distance), biomarkers (NT-proBNP and high-sensitive Troponin), and imaging markers on transthoracic echocardiography (e.g., left ventricular ejection fraction, global longitudinal strain, stroke volume index, left ventricular mass). Differences between groups for all of these variables will be analyzed with the Wilcoxon rank sum test.
All cause mortality in AS-CA with versus without CA-specific treatment | 60 months
  All-cause mortality analyzed by Cox regression analysis and Kaplan Meier estimates in AS-CA with versus without CA-specific treatment
Hospitalization for heart failure in AS-CA with versus without CA-specific treatment | 60 months
  Hospitalization for heart failure analyzed by Cox regression analysis and Kaplan Meier estimates in AS-CA with versus without CA-specific treatment
Cardiovascular mortality in AS-CA with versus without CA-specific treatment | 60 months
  Cardiovascular mortality analyzed by Cox regression analysis and Kaplan Meier estimates in AS-CA with versus without CA-specific treatment

SECONDARY OUTCOMES:
Natural history of AS-ATTR after valve replacement | 60 months
  Trajectory of morphological (left ventricular mass), functional (ejection fraction, global longitudinal strain, New York Heart Association class) and biomarker (NT-proBNP, high-sensitive Troponin) profiles. Longitudinal changes between visits will be compared using the Wilcoxon signed-rank test, McNemar's test, and the Stuart Maxwell test where appropriate.
Composite of hospitalization for heart failure and/or death in AS-CA with versus without CA-specific treatment | 60 months
  Composite of hospitalization for heart failure and/or death analyzed by Cox regression analysis and Kaplan Meier estimates in AS-CA with versus without CA-specific treatment
Heart failure hospitalzation rate in AS-CA with versus without CA-specific treatment | 36 months
  Differences in heart failure hospitalization rate, calculated as the number of heart failure hospitalizations per total person-years in AS-CA with versus without CA-specific treatment at 1 and 3 years, analyzed by the poisson model.

CONTACTS AND LOCATIONS:
Locations (2):
- Medical University of Vienna, Vienna, Austria
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nitsche C, Scully PR, Patel KP, Kammerlander AA, Koschutnik M, Dona C, Wollenweber T, Ahmed N, Thornton GD, Kelion AD, Sabharwal N, Newton JD, Ozkor M, Kennon S, Mullen M, Lloyd G, Fontana M, Hawkins PN, Pugliese F, Menezes LJ, Moon JC, Mascherbauer J, Treibel TA. Prevalence and Outcomes of Concomitant Aortic Stenosis and Cardiac Amyloidosis. J Am Coll Cardiol. 2021 Jan 19;77(2):128-139. doi: 10.1016/j.jacc.2020.11.006. Epub 2020 Nov 9. PMID 33181246
- [Result] Nitsche C, Aschauer S, Kammerlander AA, Schneider M, Poschner T, Duca F, Binder C, Koschutnik M, Stiftinger J, Goliasch G, Siller-Matula J, Winter MP, Anvari-Pirsch A, Andreas M, Geppert A, Beitzke D, Loewe C, Hacker M, Agis H, Kain R, Lang I, Bonderman D, Hengstenberg C, Mascherbauer J. Light-chain and transthyretin cardiac amyloidosis in severe aortic stenosis: prevalence, screening possibilities, and outcome. Eur J Heart Fail. 2020 Oct;22(10):1852-1862. doi: 10.1002/ejhf.1756. Epub 2020 Feb 20. PMID 32078212
- [Result] Nitsche C, Koschutnik M, Dona C, Radun R, Mascherbauer K, Kammerlander A, Heitzinger G, Dannenberg V, Spinka G, Halavina K, Winter MP, Calabretta R, Hacker M, Agis H, Rosenhek R, Bartko P, Hengstenberg C, Treibel T, Mascherbauer J, Goliasch G. Reverse Remodeling Following Valve Replacement in Coexisting Aortic Stenosis and Transthyretin Cardiac Amyloidosis. Circ Cardiovasc Imaging. 2022 Jul;15(7):e014115. doi: 10.1161/CIRCIMAGING.122.014115. Epub 2022 Jul 8. PMID 35861981
- [Result] Patel KP, Scully PR, Nitsche C, Kammerlander AA, Joy G, Thornton G, Hughes R, Williams S, Tillin T, Captur G, Chacko L, Kelion A, Sabharwal N, Newton JD, Kennon S, Ozkor M, Mullen M, Hawkins PN, Gillmore JD, Menezes L, Pugliese F, Hughes AD, Fontana M, Lloyd G, Treibel TA, Mascherbauer J, Moon JC. Impact of afterload and infiltration on coexisting aortic stenosis and transthyretin amyloidosis. Heart. 2022 Jan;108(1):67-72. doi: 10.1136/heartjnl-2021-319922. Epub 2021 Sep 8. PMID 34497140
- [Result] Scully PR, Patel KP, Saberwal B, Klotz E, Augusto JB, Thornton GD, Hughes RK, Manisty C, Lloyd G, Newton JD, Sabharwal N, Kelion A, Kennon S, Ozkor M, Mullen M, Hartman N, Cavalcante JL, Menezes LJ, Hawkins PN, Treibel TA, Moon JC, Pugliese F. Identifying Cardiac Amyloid in Aortic Stenosis: ECV Quantification by CT in TAVR Patients. JACC Cardiovasc Imaging. 2020 Oct;13(10):2177-2189. doi: 10.1016/j.jcmg.2020.05.029. Epub 2020 Aug 5. PMID 32771574
- [Result] Scully PR, Patel KP, Treibel TA, Thornton GD, Hughes RK, Chadalavada S, Katsoulis M, Hartman N, Fontana M, Pugliese F, Sabharwal N, Newton JD, Kelion A, Ozkor M, Kennon S, Mullen M, Lloyd G, Menezes LJ, Hawkins PN, Moon JC. Prevalence and outcome of dual aortic stenosis and cardiac amyloid pathology in patients referred for transcatheter aortic valve implantation. Eur Heart J. 2020 Aug 1;41(29):2759-2767. doi: 10.1093/eurheartj/ehaa170. PMID 32267922
- [Result] Treibel TA, Fontana M, Gilbertson JA, Castelletti S, White SK, Scully PR, Roberts N, Hutt DF, Rowczenio DM, Whelan CJ, Ashworth MA, Gillmore JD, Hawkins PN, Moon JC. Occult Transthyretin Cardiac Amyloid in Severe Calcific Aortic Stenosis: Prevalence and Prognosis in Patients Undergoing Surgical Aortic Valve Replacement. Circ Cardiovasc Imaging. 2016 Aug;9(8):e005066. doi: 10.1161/CIRCIMAGING.116.005066. PMID 27511979
- [Derived] Nitsche C, Dobner S, Rosenblum HR, Patel KP, Longhi S, Yilmaz A, Merlo M, Papathanasiou M, Griffin J, Oerlemans MIFJ, Gama F, Hamdan A, Kelion AD, Schuster A, Glaveckaite S, Akyol N, Porcari A, Schlender L, Capovilla T, Autherith M, Hauptmann L, Halavina K, Cavalcante JL, Fontana M, Scully PR, Moon JC, Mascherbauer J, Ristl R, Biagini E, Stortecky S, Maurer MS, Treibel TA; AS-Amyloidosis Consortium. Cardiac transthyretin amyloidosis treatment improves outcomes after aortic valve replacement for severe stenosis. Eur Heart J. 2025 Nov 21;46(44):4795-4806. doi: 10.1093/eurheartj/ehaf362. PMID 40452225